CLINICAL TRIAL: NCT04013295
Title: Prize-linked Savings Initiatives for Promoting Better Health and Economic Outcomes in Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Impact Research & Development Organization (Other); Innovations for Poverty Action (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 830084
Record Dates: First submitted 2019-07-03; First posted 2019-07-09 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: HIV/AIDS
Keywords: HIV; transactional sex; prize-linked savings; savings
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prize-linked savings intervention (Experimental): Participants in the intervention group will be assisted with opening bank accounts at the partner bank and will be eligible for monetary rewards linked to the amount they save in these project accounts. During the intervention period, information about participants' savings activities will be shared with the study team at regular intervals by the bank. Winners will learn of their prize via text message and will have their prize money deposited into their accounts. Respondents who did not win the lottery will also receive a text message, which will remind them to save.
  Interventions: Other: Prize-linked savings
- Control (No Intervention): Participants will be eligible for prizes based on the amount by which their account balance goes up in each period (e.g. for every 100 Ksh by which savings increases, participants get an entry into a lottery for monetary rewards where they have a small probability of winning a larger amount, or a larger probability of winning a smaller amount of money). This type of prize-linked savings intervention has been shown to promote savings in other settings.
  Other intervention components may include education materials to explain how the prize-linked savings incentives work and that emphasize the potential benefits of saving money. Participants in the intervention group will be encouraged to have more consideration for their future health and economic status, as this may motivate them to save more money. They will also be encouraged to consider the opportunity and health cost of their expenditures on alcohol and transactional sex and not miss the opportunity to win prizes by saving money.

INTERVENTIONS:
Other: Prize-linked savings — Participants will be eligible for prizes based on the amount by which their account balance goes up in each period (e.g. for every 100 Ksh by which savings increases, participants get an entry into a lottery for monetary rewards where they have a small probability of winning a larger amount, or a larger probability of winning a smaller amount of money). This type of prize-linked savings intervention has been shown to promote savings in other settings.
  Other intervention components may include education materials to explain how the prize-linked savings incentives work and that emphasize the potential benefits of saving money. Participants in the intervention group will be encouraged to have more consideration for their future health and economic status, as this may motivate them to save more money. They will also be encouraged to consider the opportunity and health cost of their expenditures on alcohol and transactional sex and not miss the opportunity to win prizes by saving money.
  Arms: Prize-linked savings intervention

SUMMARY:
Transactional sex is widely believed to be among the driving factors for the high HIV rates among adolescent girls and young women in Kenya. We will pilot a randomized trial among men in Kenya to assess whether prize-linked savings opportunities reduce spending on transactional sex. The project will randomize men to the savings intervention and assess changes in key economic and self-reported health outcomes over a 3-6 month period.

DETAILED DESCRIPTION:
Despite a large decline in new adult HIV infections in eastern and southern Africa from 2005-2015, progress has slowed in recent years. In particular, HIV risk among adolescent girls and young women remains high. Transactional sex, or the exchange of material support in non-commercial sexual relationships, is widely believed to be among the main driving factors for the HIV risk in this population. There is a large gap when it comes to interventions targeting men who engage in transactional sex. The proposed pilot project seeks to fill this important gap by using behavioral economic principles to promote behavior change among men.

The project will assess a novel prize-linked savings intervention designed to shift men's income away from alcohol and transactional sex and towards saving for the future. Prize-linked savings accounts offer savers a random, lottery-like payout proportional to the amount participants save, instead of traditional interest income. A number of banks, employers, and policymakers have promoted this low-cost, scalable approach to increasing savings among low-income individuals. However, there have been no assessments of whether prize-linked savings interventions can induce changes in key health-related behaviors as well. We will conduct a pilot randomized trial among men in Kenya to assess whether offering prize-linked savings opportunities leads to reduced spending on alcohol and transactional sex. The project will enroll men who in communities with high HIV risk, randomize them to the savings intervention, and assess changes in key economic and self-reported health outcomes over a 3-month period with baseline and follow-up surveys. We hypothesize that men randomized to the prize-linked savings intervention will have higher savings, lower expenditure on transactional sex, alcohol, and gambling, and lower rates of participation in risk behaviors such as transactional sex, relative to men randomized to the standard bank account control group.

ELIGIBILITY:
Inclusion Criteria:

* Resident in selected shoreline communities and their hinterlands in Siaya County, Kenya
* Male
* Age 21 years and above
* Primary or secondary occupation is fishing or transportation (i.e. motorbike taxi driver)
* Owns mobile phone
* Is willing to open savings account with a local bank and has, or is willing to obtain, the necessary documents (national identification card, Kenya Revenue authority PIN) to do so

Exclusion Criteria:

* Planning to relocate from study communities in the next 6 months
* Does not express willingness to open a savings account

Min Age: 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-18 (Actual)

PRIMARY OUTCOMES:
Increase in savings balance | Measured throughout follow-up period (approx 3 months)
  This is a binary variable equal to 1 if the respondent's savings balance increased over the study period, and zero otherwise.
Savings balance | Measured throughout follow-up period (approx 3 months)
  Total increase in savings balance over the study period (continuous measure)
Expenditures on alcohol | Recall period: past 7 days, measured in endline survey (approx 3 months after enrollment)
  Total spending on alcohol in past 7 days
Participation in and expenditures on transactional sex | Recall period: past month, measured in endline survey (approx 3 months after enrollment)
  Total spending on transactional sex in past month, and binary indicator for any spending

SECONDARY OUTCOMES:
Savings | approx 3 month follow up period
  Net increase in both the savings balance and in self-reported total savings from all sources, in each lottery period and over the entire study period
Expenditures on food | Recall period: past 7 days, measured in endline survey
  Money spent in past 7 days on food
Expenditures on non-food items | Recall period: past 7 days, measured in endline survey
  Money spent in past 7 days on all non-food items

CONTACTS AND LOCATIONS:
Overall Officials: Harsha Thirumurthy, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moscoe E, Agot K, Thirumurthy H. Effect of a Prize-Linked Savings Intervention on Savings and Healthy Behaviors Among Men in Kenya: A Randomized Clinical Trial. JAMA Netw Open. 2019 Sep 4;2(9):e1911162. doi: 10.1001/jamanetworkopen.2019.11162. PMID 31517964